CLINICAL TRIAL: NCT06671210
Title: Clinical Evaluation of Self-collected Urine Samples for the Detection of Human Papillomavirus in Males
Brief Title: Clinical Performance of Urine HPV Testing in Males
Status: Recruiting | Type: Observational
Sponsor: Peking University People's Hospital (Other)
Collaborators: Hangzhou Newhorizon Health Technology Co., Ltd. (Unknown)
Responsible Party: Principal Investigator, Zhao yongping, Principal Investigator, Peking University People's Hospital
Other Study IDs: 2024PHB118-001
Record Dates: First submitted 2024-10-30; First posted 2024-11-04 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-10

CONDITIONS: HPV; Self-sampling; Male
Keywords: urine; HPV; male

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Self-comparison
  Interventions: Device: Urine and vaginal swab self-control

INTERVENTIONS:
Device: Urine and vaginal swab self-control — Each participant provided urine and vaginal swabs for HPV testing.

SUMMARY:
Human papillomavirus (HPV) infection is one of the most prevalent viral infections of the genital tract, primarily transmitted through sexual contact. Research indicates that individuals engaging in sexual activity have a lifetime probability of HPV infection as high as 85% to 90%. While extensive and in-depth investigations have been conducted on HPV infection in women, epidemiological studies focusing on male HPV infection remain relatively scarce. Many men with HPV are asymptomatic; reports suggest that approximately 10.5% of men in China are infected with HPV, yet only about 1% exhibit related symptoms. This substantial population of asymptomatic and unaware patients poses significant challenges for the prevention and control efforts regarding HPV in China. Furthermore, evidence suggests an association between HPV infection and conditions such as condyloma acuminatum, penile intraepithelial neoplasia (PeIN), penile cancer (PA), and even infertility among male patients. In current clinical practice, detection of HPV typically involves collecting exfoliated cells from the external genitalia via swabs. The discomfort associated with this sampling method and its procedural complexity often deter many asymptomatic men from undergoing penile swab testing for HPV, resulting in low compliance rates. Self-sampling urine tests offer advantages including convenience, ease of use, painlessness, and non-invasiveness; thus they may serve as a viable alternative approach. In prior research endeavors, we successfully established a detection system utilizing female urine samples for identifying HPV presence. Consequently, this study aims to further refine this detection system to develop a stable and reliable methodology for detecting HPV using self-collected urine samples from males. Through this investigation not only do we seek to validate the feasibility of employing self-collected urine samples for detecting male HPV infections but also assess the accuracy and practicality of home-based self-testing methods among subjects-ultimately providing novel strategies for male-specific HPV detection

DETAILED DESCRIPTION:
The first part of the study aims to investigate the consistency of HPV infection between self-collected urine samples and physician-collected penile samples in male patients with genital warts, PIN and PA. Eligible subjects were enrolled, and they were first asked to collect 20-30 ml of urine by themselves, followed by physicians collecting urine samples from the urethral orifice, the surface of the external genitalia, and the surface (if any) of the lesion using urine self-collection swabs to compare the consistency of HPV infection between the two sample types. The second part of the study aims to investigate the consistency of HPV infection between urine samples of male patients and their female partners. Eligible subjects and their female partners were enrolled, and they were first asked to collect the urine sample by themselves. Urine samples were then collected from the urethral orifice and the surface of the external genitalia of the male partner by physicians using urine self-collection swabs, and a cervical swab was taken from the surface of the cervix of the female partner to compare the consistency of HPV infection between the two partners and the consistency of HPV infection between the two sample types.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years old and have had sexual experience;

  * After one year or more of regular, unprotected sexual activity without pregnancy in married couples； ③Voluntarily participate in this study after communication and sign an informed consent form.

Exclusion Criteria:

* Samples that cannot obtain valid nucleic acid test results, including but not limited to samples with human errors in clinical trial testing process or samples with insufficient volume to complete a valid test; ② Incomplete demographic information and laboratory test related information of the subjects.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult men who meet the inclusion criteria, or infertile couples, who are willing to participate in a clinical trial and seek treatment at the Dermatology and Reproductive Medicine Department of Peking University People's Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-11-04 (Actual); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Compare the test results of the candidate reagent for HPV detection on appropriate urine samples from the same male subject with the results of the marketed HPV nucleic acid detection products on external genital samples of the subject. | 12weeks

SECONDARY OUTCOMES:
Compare the consistency of HPV nucleic acid in urine samples of male subjects and their spouses to explore the feasibility of using the under-evaluation reagent for couples' joint testing with suitable urine samples. | 8weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Garland SM, Kjaer SK, Munoz N, Block SL, Brown DR, DiNubile MJ, Lindsay BR, Kuter BJ, Perez G, Dominiak-Felden G, Saah AJ, Drury R, Das R, Velicer C. Impact and Effectiveness of the Quadrivalent Human Papillomavirus Vaccine: A Systematic Review of 10 Years of Real-world Experience. Clin Infect Dis. 2016 Aug 15;63(4):519-27. doi: 10.1093/cid/ciw354. Epub 2016 May 26. PMID 27230391
- [Background] Smits PH, Bakker R, Jong E, Mulder JW, Meenhorst PL, Kleter B, van Doorn LJ, Quint WG. High prevalence of human papillomavirus infections in urine samples from human immunodeficiency virus-infected men. J Clin Microbiol. 2005 Dec;43(12):5936-9. doi: 10.1128/JCM.43.12.5936-5939.2005. PMID 16333078
- [Background] Wu H, Tong X, Wang L, Huang Y, Zhang L. HPV vaccine information, knowledge, attitude, and recommendation intention among male college students in China. Hum Vaccin Immunother. 2023 Aug 1;19(2):2228163. doi: 10.1080/21645515.2023.2228163. PMID 37389484
- [Background] Chesson HW, Dunne EF, Hariri S, Markowitz LE. The estimated lifetime probability of acquiring human papillomavirus in the United States. Sex Transm Dis. 2014 Nov;41(11):660-4. doi: 10.1097/OLQ.0000000000000193. PMID 25299412